CLINICAL TRIAL: NCT07097688
Title: Regenerative Endodontic Treatment Using Sodium Hexametaphosphate (SHMP) For Necrotic Immature Permanent Anterior Teeth: In Vivo And In Vitro Study
Brief Title: Regenerative Endodontic Treatment Using Sodium Hexametaphosphate (SHMP) For Necrotic Immature Permanent Anterior Teeth
Acronym: Regeneration
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Ahmad Elheeny (Other)
Responsible Party: Sponsor-Investigator, Ahmad Elheeny, Assistant professor of Pediatric and Community Dentistry, Faculty of Dentistry, Minia University, Minia University
Organization: Minia University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Regenerative Endodontic Treatm
Record Dates: First submitted 2025-07-01; First posted 2025-07-31 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-07

CONDITIONS: Regenerative Inflammation
Keywords: regeneration ,immature teeth ,sodiumhexametaphosphate ,MTA
MeSH Terms: interventions — sodium polymetaphosphate

STUDY DESIGN:
Intervention Model Description: Included patients will be randomized into one of the study groups. Randomization will be performed using a computer-generated block randomization system (Microsoft office excel, 2007).
  Concealment, A plan of management will be sealed in closed envelops, numbered according to the randomization tables.
  Packing, sealing and numbering will all be performed by a neutral health care provider other than the investigator
Who Masked: Investigator
Masking Description: -Included patients will be randomized into one of the study groups. Randomization will be performed using a computer-generated block randomization system (Microsoft office excel, 2007).
  Concealment, A plan of management will be sealed in closed envelops, numbered according to the randomization tables.
  Packing, sealing and numbering will all be performed by a neutral health care provider other than the investigator.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Sodium Hexametaphosphate (Active Comparator): dental material
  Interventions: Biological: Sodium Hexametaphosphate (SHMP) Inorganic polyphosphates (poly[P]) are linear polymers of orthophosphate (Pi) residues linked by energy-rich phosphoranhydride bonds, Ithas multiple physiological funct
- Mineral Trio oxide Aggregate (No Intervention): dental biological and compatible material

INTERVENTIONS:
Biological: Sodium Hexametaphosphate (SHMP) Inorganic polyphosphates (poly[P]) are linear polymers of orthophosphate (Pi) residues linked by energy-rich phosphoranhydride bonds, Ithas multiple physiological funct — The study will be with two parallel arms (1:1 allocation ratio). The sample size per group will be calculated according to the following equation for binary outcomes; N = (Zα/2 + Zβ) 2 ×p1(1 - p1) + p2(1 - p2)/δ 2 so the minimal sample size for an equal size clinical trial is 27teeth in each group. We will recruit 30 teeth in each group for possible attrition
  Arms: Sodium Hexametaphosphate

SUMMARY:
evaluate clinically and radiographically regenerative potential of sodium hexametaphosphate (SHMP) on stem cells from the apical papilla for 18-month randomized controlled trial

DETAILED DESCRIPTION:
7 to 11 years old will be selected with no sex predilection for the study from out patients of Pediatric and Community Dentistry Department, Minia University, according to the following eligibility criteria and evaluate clinically and radiographically regenerative potential of sodium hexametaphosphate (SHMP) on stem cells from the apical papilla for 18-month randomized controlled trial

ELIGIBILITY:
Inclusion Criteria:

Presence of necrotic anterior immature teeth. Parents accepting the treatment modality.History, clinical and radiographic examination reveals absence of pulp vitality Patient abruptly health

Exclusion Criteria:

Tooth mobility. Children who will not comply to recall program. Teeth with history of recurrent periapical pathosis. Hypersensitivity to any material used.

Ages: 7 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2025-06-29 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
Normal responses to percussion, palpation, and normal pocket probing depths, and a positive response to pulp test | one year
  pulp sensibility test
Absence of signs and symptoms of pain, absence of mobility or periapical lesion | one year
  PALS scale

CONTACTS AND LOCATIONS:
Overall Officials: minia university, Principal Investigator — minia university faculty of dentistry
Locations (1):
- Faculty of Dentistry, Minya, Egypt

IPD SHARING:
Plan to Share IPD: No
All patients and their caregivers will be informed in an easy detailed manner about the treatment procedures, expected outcome of the current treatment, possibility of any complications and assuring them to presence of plan B in case of any complication. Verbal assent will be obtained from all children who will accept participation in the study, Parents will sign an informed consent laid down by ethical committee of Faculty of Dentistry / Minia University